CLINICAL TRIAL: NCT00438425
Title: Assessment of the Practical Application, Acceptability and Effectiveness of a Portfolio Diet in Reducing Serum Cholesterol
Brief Title: Portfolio 5 - Multicentre Dietary Advice on Serum Lipids in Hyperlipidemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Loblaw Companies Limited (Industry); Solae, LLC (Industry); Unilever R&D (Industry)
Responsible Party: Principal Investigator, David Jenkins, Principle Investigator, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REB 04-056c; CIHR RCT#: 68767
Record Dates: First submitted 2007-02-21; First posted 2007-02-22 (Estimated); Last update posted 2018-10-15 (Actual); Status verified 2018-10

CONDITIONS: Hyperlipidemia; Cardiovascular Disease
Keywords: Hyperlipidemia; Hypercholesterolemia; Dietary modification; Portfolio
MeSH Terms: conditions — Hyperlipidemias; Cardiovascular Diseases; Hypercholesterolemia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Intensive Portfolio (Experimental): The portfolio dietary advice will conform to current therapeutic diets appropriate for hypercholesterolemic subjects (<7% of energy saturated fat, <200 mg/d cholesterol) plus the combination of viscous fibers, soy protein, plant sterols and nuts. The portfolio diet plan will include foods which contribute 9.8 g/1000 kcal viscous fiber as B-glucan (oats, barley, oat bran breads and soups) and psylliium (cereal), 0.94 g plant sterol/1000 kcal diet (in sterol margarine), 22.5 g soy protein/1000 kcal (soy burgers, dogs, links, other meat analogues, milks, yogurts and cheese) and 22.5 g nuts/1000 kcal. Participants received 7 visits during a 6-month period with the study dietitian.
  Interventions: Dietary Supplement: Dietary Portfolio - Intensive
- Routine Portfolio (Experimental): The portfolio dietary advice will conform to current therapeutic diets appropriate for hypercholesterolemic subjects (<7% of energy saturated fat, <200 mg/d cholesterol) plus the combination of viscous fibers, soy protein, plant sterols and nuts. The portfolio diet plan will include foods which contribute 9.8 g/1000 kcal viscous fiber as B-glucan (oats, barley, oat bran breads and soups) and psylliium (cereal), 0.94 g plant sterol/1000 kcal diet (in sterol margarine), 22.5 g soy protein/1000 kcal (soy burgers, dogs, links, other meat analogues, milks, yogurts and cheese) and 22.5 g nuts/1000 kcal. Participants received 2 visits during a 6-month period with the study dietitian.
  Interventions: Dietary Supplement: Dietary Portfolio - Routine
- Control (Active Comparator): Advice focused on low-fat dairy and whole grain cereals together with fruit and vegetables as part of a low fat vegetarian diet, and avoidance of the specific portfolio components.
  Interventions: Dietary Supplement: Control (low saturated fat therapeutic diet)

INTERVENTIONS:
Dietary Supplement: Dietary Portfolio - Intensive — Dietitians advised participants to consume the following therapeutic diet components (<7% of energy saturated fat, <200 mg/d cholesterol) plus the combination of viscous fibers, soy protein, plant sterols and nuts. The portfolio diet plan will include foods which contribute 9.8 g/1000 kcal viscous fiber as B-glucan (oats, barley, oat bran breads and soups) and psylliium (cereal), 0.94 g plant sterol/1000 kcal diet (in sterol margarine), 22.5 g soy protein/1000 kcal (soy burgers, dogs, links, other meat analogues, milks, yogurts and cheese) and 22.5 g nuts/1000 kcal as part of a low fat vegetarian diet. Participants received 7 visits during a 6-month period with the study dietitian.
  Arms: Intensive Portfolio
Dietary Supplement: Dietary Portfolio - Routine — Dietitians advised participants to consume the following therapeutic diet components (<7% of energy saturated fat, <200 mg/d cholesterol) plus the combination of viscous fibers, soy protein, plant sterols and nuts. The portfolio diet plan will include foods which contribute 9.8 g/1000 kcal viscous fiber as B-glucan (oats, barley, oat bran breads and soups) and psylliium (cereal), 0.94 g plant sterol/1000 kcal diet (in sterol margarine), 22.5 g soy protein/1000 kcal (soy burgers, dogs, links, other meat analogues, milks, yogurts and cheese) and 22.5 g nuts/1000 kcal as part of a low fat vegetarian diet. Participants received 2 visits during a 6-month period with the study dietitian.
  Arms: Routine Portfolio
Dietary Supplement: Control (low saturated fat therapeutic diet) — Dietitians advised participants to consume the following therapeutic diet components (<7% of energy saturated fat, <200 mg/d cholesterol) with a focus on low-fat dairy and whole grain cereals together with fruit and vegetables as part of a low fat vegetarian diet, and avoidance of the specific portfolio components.
  Arms: Control

SUMMARY:
The purpose of this trial is to re-evaluate the potential role of diet in modulating cardiovascular risk factors. If potent lipid-lowering effects through novel dietary interventions can be demonstrated, then diet may again be seen as providing an alternative to drug therapy in the primary prevention of cardiovascular disease.

Aims:

* To determine the percentage of lipid clinic attendees interested in making a serious dietary change.
* To determine the extent to which a self selected dietary portfolio combining viscous fiber foods (oat & barley β-glucan, psyllium, etc.), soy and vegetable protein foods (soy milk, soy meat analogues and almonds) and plant sterols (sterol margarine) in the same diet be significantly more effective in reducing LDL-cholesterol and other markers of cardiovascular disease risk than conventional dietary advice.
* To determine whether this effect can be maximized by more frequent follow-up, and what, if any, would be the relationship between dietary compliance and reduction in LDL-C.

DETAILED DESCRIPTION:
This is a randomized parallel study with three experimental arms of 6 months duration to estimate the effect of the portfolio diet under real world conditions at two levels of advice intensity. Every effort will be made to obtain study blood samples and other data from all subjects at the designated times regardless of compliance with the dietary aspects of the study protocol. All subjects will be used in the intent-to-treat analysis.

Four Canadian Centers will be involved: Vancouver, Toronto, Manitoba and Quebec City. The study will be partially blinded. The investigators and technical staff will be blinded but the dietitians and the patients will not be, owing to the differences in taste and appearance of the study foods. The blinding of physicians at clinic visits is likely to be difficult due to the requirement to ask questions related to diet. All patients referred to the four collaborating clinics will be asked whether they would be prepared to modify their diet if that may mean they might lower their blood cholesterol without the use of drugs. Those who checked the box for "No" or "only modest dietary change" would not be considered further. Those who checked the box for "significant" or "radical dietary change" would be invited to participate, providing they are not at high risk (<20% 10 yr risk) of CHD and were within 30% of their target LDL-C concentrations according to current Canadian Working Group recommendations i.e., those who would normally be considered for a preliminary test of diet. The three groups would be randomized to either a low saturated fat, low cholesterol diet (Step 2) or a portfolio diet both given as routine clinical advice at week zero with follow up at 3 and 6 months or more intensive advice reinforced (intensive portfolio) at clinic visits at 2, 4, 8, 12, 16 and 20 weeks. In the routine portfolio, the advice will therefore consist of two half hour sessions with the dietitian (0 and 12 weeks), compared to seven for the intensive portfolio (0, 2, 4, 8, 12, 16 and 20 weeks). Prior to starting each diet the nature of the diet will be explained to the participants and instruction on achieving diet goals will be given. Follow-up visits will be used to go over the subjects' diet record, which they have recorded over the previous 7 days, and reinforce the original dietary advice. The intensive portfolio participants will therefore receive five additional instructional and assessment follow up visits during the course of the study.

Trial treatments: The portfolio dietary advice will conform to current therapeutic diets appropriate for hypercholesterolemic subjects (<7% of energy saturated fat, <200 mg/d cholesterol) plus the combination of viscous fibers, soy protein, plant sterols and almonds. The portfolio diet plan will include foods which contribute 8 g/1000 kcal viscous fiber as β-glucan (oats, barley, oat bran breads and soups) and psyllium (cereal), 1 g plant sterol/1000 kcal diet (in sterol margarine), 22 g soy protein/1000 kcal (soy burgers, dogs, links, other meat analogues, milks, yogurts and cheese) and 22 g almonds/1000 kcal. The Step 2 therapeutic diet will encourage a similar macronutrient profile through the use of cereal fibers and whole grains. All diets will emphasize fruit and vegetable intakes (5-10 servings/d) according to current recommendations. Participants will be instructed on how to select and follow these diets and will be provided with only the margarine component of the portfolio and Step 2 therapeutic diets. The Step 2 therapeutic diet group will be encouraged to follow a diet of whole grain foods (brown rice, whole wheat breads, muffins and breakfast cereals), low saturated fat meat and dairy foods with a control margarine. The degree to which the portfolio diet can be made effective after routine instruction compared to more intensive instruction is the key issue in this study.

Duration of Subject participation and sequence and duration of all trial periods: Subject participation will start with the screening visit followed by a week minus 2 visit 4 to 6 weeks later. The week minus 2 visit will be followed by week 0 visit. Study duration is for 6 months, after which participants have the option of continuing for another 6 months.

Diets will be self-selected, low-fat, low-cholesterol, NCEP Step 2 diets (<7% saturated fats, <200 mg dietary cholesterol/d). The test and control margarines will be provided free. The oat bran bread will be provided at cost. The control diet will encourage a low saturated fat intake (<7%) by the use of low fat dairy products and egg substitutes (Fleischmann's egg beaters). Fiber will be increased to 17 g/1000 kcal recommending insoluble cereal fiber and whole meal or whole grain flour cereal products which are lipid neutral but conform to current diet guidelines for fiber intake and appear to offer protection from CHD. This will ensure equal total fiber intake on the NCEP and Portfolio diet. The control margarine (45 g/d) will have the same fatty acid composition as the test margarine. The Portfolio treatment diet will have a similar fatty acid and macronutrient profile to the control treatment diet. Low-fat Dairy and egg protein sources will be replaced with soy (approximately 45 g/d) protein. Foods will include soy dairy foods (milks, yogurts & cheese), and meat analogues made from soy isolate (dogs and burgers etc) and tofu products. The fiber will include at least 15 g viscous fiber daily from oats, barley, dried beans, peas, lentils and psyllium cereal. Plant sterols (1g/1000 kcal diet) up to 3g/day will be recommended from the test margarine provided which will be consumed up to a quantity of 40 g/day. A control margarine in the same quantity (25-40 g/d) will be provided to the participants in the control group. Almonds (22g/1000 kcal), the FDA recommended dose for cholesterol reduction) will also be included in the diet. The protein and fiber components will be individualized as much as possible to achieve study goals while satisfying individual preferences. The portfolio diet will be prescribed at two levels of reinforcement. In one portfolio cohort, the advice will be general and provided on 2 occasions over a 6 month period. For the second portfolio cohort, the advice will be much more intensive and provided on 7 occasions (total of 8 visits) over a 6 month period. Participants in the control and less intensive portfolio treatment groups will be seen at weeks 0, 12, 24 and optionally at 36 and 52 weeks. While participants in the intensive portfolio treatment group will be seen at two-weekly intervals for the first month and then monthly for the next five months (with a final visit at 6 months) and at two monthly intervals thereafter (if study is extended to 12 months) to ensure the diet plan is acceptable. Participants, in the intensive advice group, will be provided with self-taring scales on which to weigh all food to be consumed.

ELIGIBILITY:
Inclusion Criteria:

* Men over the age of 21 years and postmenopausal women with mild-to-moderate hypercholesterolaemia, for whom cholesterol lowering medications are being considered
* Body mass index <35 kg/m2.
* Treated by diet
* Alcohol intake < 14 drinks per week.
* Fasting plasma triglyceride (TG) concentration <4.5 mmol/l.
* Fasting plasma LDL cholesterol concentration > 4.1 mmol/l at diagnosis or within 30% of their target levels based on risk
* Patients with previous adverse effects on statins (e.g. muscle pains) will also be accepted if the physician responsible for their care considers it appropriate.
* Individuals who prior to cholesterol lowering therapy or after discontinuing cholesterol lowering therapy are within 30% of their treatment LDL-C goals may be permitted to enter the study with the approval of their responsible physician.
* Fit individuals who have had a myocardial infarction or cardiac bypass surgery in the past will not be excluded. Their responsible physician will be asked to provide a letter confirming their suitability for the study.

Exclusion Criteria:

* Premenopausal women will be excluded due to the fluctuation of blood lipids during the menstrual cycle.
* Patients will be excluded if they are taking cholesterol medications at the start of the study. However, with their physician's approval, those who wish to join but are already taking cholesterol-lowering medications may join the study providing the medications are stopped for one month before starting the study and throughout the study.
* Patients will be excluded if they are taking cholesterol lowering natural health products such as psyllium, red yeast rice, cholest, polycosanol etc. However, they will be allowed to join the study if they are willing to discontinue these products at least 2 weeks before the start of the study and throughout the study.
* Patients with uncontrolled high blood pressure will be excluded. The cut off for raised blood pressure has been taken as > 140/90mmHg. Patients with systolic blood pressure between 140-150mmHg and diastolic blood pressure between 90-95mmHg may be accepted, since we have found that on the diet their blood pressures tend to be lowered into the acceptable range. For patients in the above normal range (as above), a letter will be required from the physician responsible for their care. Patients will be excluded if they change the type or dose of their blood pressure treatment during the study.
* Patients will be excluded if they are judged as having a likelihood of being non-compliant with instructions for whatever reason. Those with low compliance to lipid-lowering therapy will not be selected.
* Patients will be excluded if they have evidence or history of diabetes, renal disease, liver disease or gastrointestinal disease. Patients will be excluded if they have gross xanthoma or advanced premature cardiovascular disease since this group may include hyper-absorbers of plant sterols.
* Individuals predisposed to hemorrhagic stroke (on the basis of untreated raised blood pressure) will be excluded.
* Patients will be excluded from the study if they have a history of any form of cancer apart from non melanoma skin cancer or are considered at high risk for cancer. However, if such patients wish to join the study, we would like them to obtain the approval of their oncologist or responsible physician prior to enrollment in the study. If the study oncologist does not believe it is safe to enroll the participant, the patient will be excluded from the study.

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 351 (Actual)
Dates: Start 2007-06-25 (Actual); Primary Completion 2009-09-30 (Actual); Study Completion 2010-03-31 (Actual)

PRIMARY OUTCOMES:
Primary Outcome Measures Described Below | December 2011
  Plasma LDL-C concentrations

SECONDARY OUTCOMES:
Secondary Outcome Measures Described Below | January 2016 (anticipated)
  Total-C:HDL-C ratio, total-C, triglycerides, HDL-C, apolipoproteins A-1 and B, LDL particle size, oxidized LDL (conjugated dienes), Lp(a), homocysteine, C-reactive protein, glucose and insulin, waist circumference, blood pressure, diet records focusing on the intake of saturated fat and the amounts of the four key dietary components of the portfolio diet (viscous fibers, soy proteins, plant sterols, and almonds). Urinary urea, creatinine, and minerals.

OTHER OUTCOMES:
Tertiary Outcome Measures Described Below | January 2016 (anticipated)
  Plasma and red cell membrane sterols and red cell membrane sterols and red cell membrane integrity (erythrocyte fragility).

CONTACTS AND LOCATIONS:
Overall Officials: David J.A. Jenkins, MD, PhD, Principal Investigator — University of Toronto, St. Michael's Hospital; Cyril W.C. Kendall, PhD, Study Director — University of Toronto, St. Michael's Hospital; Dorothea Faulkner, PhD, Study Chair — Unity Health Toronto; Benoit Lamarche, PhD, Study Director — Lipid Research Clinic & Institute on Nutraceuticals and Functional Foods, Laval University; Peter Jones, PhD, Study Director — Richardson Centre for Functional Foods and Nutraceuticals, University of Manitoba; Jiri Frohlich, MD, Study Director — Healthy Heart Program, St. Paul's Hospital, Vancouver BC.; Jay Silverberg, MD, Study Director — Sunnybrooke Health Science Centre
Locations (5):
- Canada (5):
  - Healthy Heart Program, St. Paul's Hospital, Vancouver, British Columbia
  - Richardson Centre for Functional Foods and Nutraceuticals, University of Manitoba, Winnipeg, Manitoba
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Institute on Nutraceuticals and Functional Foods and the Lipid Research Center, Laval University Hospital Research Center, Québec, Quebec

REFERENCES:
- [Background] Jenkins DJ, Kendall CW, Faulkner DA, Nguyen T, Kemp T, Marchie A, Wong JM, de Souza R, Emam A, Vidgen E, Trautwein EA, Lapsley KG, Holmes C, Josse RG, Leiter LA, Connelly PW, Singer W. Assessment of the longer-term effects of a dietary portfolio of cholesterol-lowering foods in hypercholesterolemia. Am J Clin Nutr. 2006 Mar;83(3):582-91. doi: 10.1093/ajcn.83.3.582. PMID 16522904
- [Background] Jenkins DJ, Kendall CW, Marchie A, Faulkner DA, Josse AR, Wong JM, de Souza R, Emam A, Parker TL, Li TJ, Josse RG, Leiter LA, Singer W, Connelly PW. Direct comparison of dietary portfolio vs statin on C-reactive protein. Eur J Clin Nutr. 2005 Jul;59(7):851-60. doi: 10.1038/sj.ejcn.1602152. PMID 15900306
- [Background] Jones PJ, Raeini-Sarjaz M, Jenkins DJ, Kendall CW, Vidgen E, Trautwein EA, Lapsley KG, Marchie A, Cunnane SC, Connelly PW. Effects of a diet high in plant sterols, vegetable proteins, and viscous fibers (dietary portfolio) on circulating sterol levels and red cell fragility in hypercholesterolemic subjects. Lipids. 2005 Feb;40(2):169-74. doi: 10.1007/s11745-005-1372-6. PMID 15884765
- [Background] Jenkins DJ, Kendall CW, Marchie A, Faulkner DA, Wong JM, de Souza R, Emam A, Parker TL, Vidgen E, Trautwein EA, Lapsley KG, Josse RG, Leiter LA, Singer W, Connelly PW. Direct comparison of a dietary portfolio of cholesterol-lowering foods with a statin in hypercholesterolemic participants. Am J Clin Nutr. 2005 Feb;81(2):380-7. doi: 10.1093/ajcn.81.2.380. PMID 15699225
- [Background] Lamarche B, Desroches S, Jenkins DJ, Kendall CW, Marchie A, Faulkner D, Vidgen E, Lapsley KG, Trautwein EA, Parker TL, Josse RG, Leiter LA, Connelly PW. Combined effects of a dietary portfolio of plant sterols, vegetable protein, viscous fibre and almonds on LDL particle size. Br J Nutr. 2004 Oct;92(4):657-63. doi: 10.1079/bjn20041241. PMID 15522135
- [Background] Jenkins DJ, Kendall CW, Marchie A, Faulkner DA, Wong JM, de Souza R, Emam A, Parker TL, Vidgen E, Lapsley KG, Trautwein EA, Josse RG, Leiter LA, Connelly PW. Effects of a dietary portfolio of cholesterol-lowering foods vs lovastatin on serum lipids and C-reactive protein. JAMA. 2003 Jul 23;290(4):502-10. doi: 10.1001/jama.290.4.502. PMID 12876093
- [Background] Jenkins DJ, Kendall CW, Faulkner D, Vidgen E, Trautwein EA, Parker TL, Marchie A, Koumbridis G, Lapsley KG, Josse RG, Leiter LA, Connelly PW. A dietary portfolio approach to cholesterol reduction: combined effects of plant sterols, vegetable proteins, and viscous fibers in hypercholesterolemia. Metabolism. 2002 Dec;51(12):1596-604. doi: 10.1053/meta.2002.35578. PMID 12489074
- [Derived] Hooper L, Abdelhamid AS, Jimoh OF, Bunn D, Skeaff CM. Effects of total fat intake on body fatness in adults. Cochrane Database Syst Rev. 2020 Jun 1;6(6):CD013636. doi: 10.1002/14651858.CD013636. PMID 32476140
- [Derived] Jenkins DJ, Jones PJ, Frohlich J, Lamarche B, Ireland C, Nishi SK, Srichaikul K, Galange P, Pellini C, Faulkner D, de Souza RJ, Sievenpiper JL, Mirrahimi A, Jayalath VH, Augustin LS, Bashyam B, Leiter LA, Josse R, Couture P, Ramprasath V, Kendall CW. The effect of a dietary portfolio compared to a DASH-type diet on blood pressure. Nutr Metab Cardiovasc Dis. 2015 Dec;25(12):1132-9. doi: 10.1016/j.numecd.2015.08.006. Epub 2015 Nov 6. PMID 26552742
- [Derived] Ramprasath VR, Jenkins DJ, Lamarche B, Kendall CW, Faulkner D, Cermakova L, Couture P, Ireland C, Abdulnour S, Patel D, Bashyam B, Srichaikul K, de Souza RJ, Vidgen E, Josse RG, Leiter LA, Connelly PW, Frohlich J, Jones PJ. Consumption of a dietary portfolio of cholesterol lowering foods improves blood lipids without affecting concentrations of fat soluble compounds. Nutr J. 2014 Oct 18;13:101. doi: 10.1186/1475-2891-13-101. PMID 25326876
- [Derived] Jenkins DJ, Jones PJ, Lamarche B, Kendall CW, Faulkner D, Cermakova L, Gigleux I, Ramprasath V, de Souza R, Ireland C, Patel D, Srichaikul K, Abdulnour S, Bashyam B, Collier C, Hoshizaki S, Josse RG, Leiter LA, Connelly PW, Frohlich J. Effect of a dietary portfolio of cholesterol-lowering foods given at 2 levels of intensity of dietary advice on serum lipids in hyperlipidemia: a randomized controlled trial. JAMA. 2011 Aug 24;306(8):831-9. doi: 10.1001/jama.2011.1202. PMID 21862744